CLINICAL TRIAL: NCT00975767
Title: A Phase I/II Study of MGCD265 in Combination With Erlotinib or Docetaxel in Subjects With Advanced Malignancies and in Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of MGCD265 Given With Erlotinib or Docetaxel in Subjects With Advanced Malignancies or Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a need for a reformulation of the study drug. Phase 1 completed, no patients enrolled in Phase 2.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 265-103
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Malignancies, Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGCD265+erlotinib (Experimental)
  Interventions: Drug: MGCD265+erlotinib
- MGCD265+docetaxel (Experimental)
  Interventions: Drug: MGCD265+docetaxel

INTERVENTIONS:
Drug: MGCD265+erlotinib — MGCD265 and erlotinib administered daily
  Arms: MGCD265+erlotinib
Drug: MGCD265+docetaxel — MGCD265 administered daily; docetaxel administered once every 3 weeks
  Arms: MGCD265+docetaxel

SUMMARY:
The main purpose of this study is to assess the safety profile of MGCD265 when administered in combination with the marketed anticancer drugs erlotinib and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Part 1:

  * Patients with advanced metastatic or unresectable solid malignancy that is refractory to standard therapy and/or existing therapies.
  * Evaluable disease.
  * Documented progressive disease during or following most recent treatment regimen.
  * Adequate hepatic parameters.
  * Age ≥18 years.
  * Life expectancy greater than 3 months.
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Adequate renal function.
  * Adequate bone marrow function.
  * Capable of understanding and complying with the protocol and written informed consent.
  * Negative pregnancy test for women of childbearing potential.
  * Use of adequate contraception as needed.
  * Subjects consenting to optional fresh biopsies, must not require concurrent anticoagulation medication.
* Part 2:

  * Histologically or cytologically confirmed advanced Stage 3b or 4 NSCLC.
  * Measurable disease per RECIST.
  * At least one prior chemotherapy regimen for advanced disease.
  * No prior erlotinib or docetaxel therapy.
  * Documented progressive disease during or following most recent treatment regimen.
  * Adequate hepatic parameters.
  * Age ≥18 years.
  * Life expectancy greater than 3 months.
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Adequate renal function.
  * Adequate bone marrow function.
  * Capable of understanding and complying with the protocol and written informed consent.
  * Negative pregnancy test for women of childbearing potential.
  * Use of adequate contraception as needed.

Exclusion Criteria:

* Recent anticancer treatment.
* Prior treatment with an investigational cmet inhibitor or HCF inhibitor or antibody.
* Uncontrolled concurrent illness.
* History of bleeding diathesis or coagulopathy.
* History of stroke or transient ischemic attack.
* History of a cardiovascular illness.
* QT interval corrected for heart rate (QTc) >470 msec.
* Left ventricular ejection fraction (LVEF) <50%.
* Immunocompromised subjects.
* Lack of recovery to grade ≤1 from significant adverse events due to antineoplastic agents, investigational drugs, or other medications administered prior to study enrollment.
* Symptomatic or uncontrolled brain metastases requiring current treatment.
* Active gastrointestinal conditions or a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess.
* History of other malignancy treated with curative intent within the 5 previous years.
* Lung tumor lesions with increased likelihood of bleeding.
* History of major surgery within 28 days of first receipt of study drug.
* History of autologous bone marrow transplant (BMT) within the previous five years, or subjects with organ transplants or allogeneic BMT.
* Nursing or pregnant women; female subjects of childbearing potential must have a negative pregnancy test at screening.
* Unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with proper absorption of oral drugs.
* Any other condition or finding that in the opinion of the Investigator or Medical Monitor may render the subject at excessive risk for treatment complications or may render difficult the evaluation of treatment response.
* Allergy or hypersensitivity to components of either the MGCD265, erlotinib or docetaxel formulations (depending on the group that the subject is assigned to).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Phase I: Safety profile (including maximum tolerated dose and dose limiting toxicities) | 1 year
Phase II: Antitumor activity of MGCD265+erlotinib and MGCD265+docetaxel | 1 year

SECONDARY OUTCOMES:
Phase I: Pharmacokinetic profiles of MGCD265+erlotinib and MGCD265+docetaxel | 2 months
Phase I and Phase II: Pharmacodynamic profiles of MGCD265+erlotinib and MGCD265+docetaxel | 1 year
Phase I: Antitumor activity of MGCD265+erlotinib and MGCD265+docetaxel. | 1 year
Phase II: Safety profile of MGCD265+erlotinib and MGCD265+docetaxel; | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Tassell, Study Director — MethylGene Inc.
Locations (5):
- United States (5):
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

REFERENCES:
- [Derived] Patnaik A, Gadgeel S, Papadopoulos KP, Rasco DW, Haas NB, Der-Torossian H, Faltaos D, Potvin D, Tassell V, Tawashi M, Chao R, O'Dwyer PJ. Phase I Study of Glesatinib (MGCD265) in Combination with Erlotinib or Docetaxel in Patients with Advanced Solid Tumors. Target Oncol. 2022 Mar;17(2):125-138. doi: 10.1007/s11523-022-00875-0. Epub 2022 Mar 28. PMID 35347559